CLINICAL TRIAL: NCT05899335
Title: Feasibility Study of a Mobile Health App for Symptom Monitoring in People With Chronic Pancreatitis: The SmartCP Study
Brief Title: Feasibility Study of a Mobile Health App for Symptom Monitoring in People With Chronic Pancreatitis
Acronym: SmartCP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Sinead Duggan, Principal Investigator, University of Dublin, Trinity College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCP001
Record Dates: First submitted 2023-05-08; First posted 2023-06-12 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SmartCP app (Experimental): The SmartCP app is provided to patients to assist in the management of chronic pancreatitis for 16 weeks
  Interventions: Device: SmartCP (mobile phone app)

INTERVENTIONS:
Device: SmartCP (mobile phone app) — As described
  Other Names: Co-designed with MyPatientSpace https://www.mypatientspace.com

SUMMARY:
Patients with chronic pancreatitis suffer from constant debilitating symptoms. They have complex needs and require specialist, multi-disciplinary care. The investigators have developed a mobile phone app for patients with chronic pancreatitis, called the SmartCP app - the first app of its kind for this patient group.

What is SmartCP? SmartCP is an app that allows patients to log daily symptoms, diet, and physical activity for review at clinic. It creates a red-alert for action if there are worsening symptoms. A Monthly-Check-In feature looks for symptoms of new diabetes or pancreatic cancer. SmartCP provides education on every aspect of pancreatitis, as well as contact information for the clinical team and for important pancreatitis resources. To develop SmartCP, the investigators established a multidisciplinary steering committee.

The study The investigators aim to conduct a feasibility study to determine if the SmartCP app is feasible in the management of patients with chronic pancreatitis, complementing current specialist healthcare. Specifically, they will investigate acceptability, retention, incidents, resources, app user statistics, as well as investigating the occurrence of crisis events, symptoms, escalating symptoms, new diagnoses of diabetes or pancreatic cancer, and the use of communication and education features.

DETAILED DESCRIPTION:
Background and rationale Chronic pancreatitis is an inherently complex disease requiring coordinated, multidisciplinary care. Patients suffer from constant, distressing, adverse symptoms including abdominal pain, steatorrhoea, bloating, wind, cramping, and fatigue - making it difficult to eat a normal or sufficient diet. They develop vitamin deficiencies, osteoporosis, and a difficult-to-manage diabetes subgroup (type 3c diabetes). There is no effective medical/surgical treatment, and the disease is progressive and incurable. The mainstay of treatment is diet, supplementation, and pancreatic enzyme replacement therapy- which helps patients to digest and absorb their food, alleviating symptoms somewhat. Contrary to perceptions, half of patients (or fewer) have an alcohol related aetiology.

The investigators run several out-patient clinics for chronic pancreatitis including medical-led, nurse-specialist led, and type 3c diabetes clinics. A nurse specialist deal with 3-5 crisis phonically daily, each lasting up to 30mins. Patients have frequent urgent clinic attendance, A&E, and hospital admissions.

What is the intervention? A steering group designed and developed the SmartCP mobile phone app during 2022 with the support of a government innovation grant. SmartCP consists of a symptom tracker, diet/physical activity log, alert system for escalating symptoms, quality of life assessment, red-flag alerts for diabetes/pancreatic cancer, educational content, push notifications and messaging function.

Overall aim of the study To conduct a study to determine if SmartCP is feasible in the management patients with chronic pancreatitis, complementing current specialist clinical care.

Design A single-arm, unblinded, feasibility study, with an uncontrolled, within-group baseline and post-intervention (16-week) design, with an embedded quantitative and qualitative process evaluation. Participants will receive the intervention for 16 weeks, supplementing usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Ireland
* Can read/write in English
* Have daily access to compatible smartphone
* Have daily access to home internet

Exclusion Criteria:

* Reside outside Ireland
* Acutely unwell
* Has multi-morbidity
* Is current inpatient
* Has prognosis <6months
* Has pancreatic cancer
* Is <18 years
* Has no access to compatible smartphone
* Has no access to home internet
* Cannot read/write in English
* Is unwilling/unable to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Recruitment | 16 weeks
  The number of participants that are recruited versus the number eligible for recruitment
Feasibility: Acceptability | 16 weeks
  Acceptability of intervention (Telehealth Usability Questionnaire; 21 questions with scale of 1 to 7 for each question, with higher scores indicating more positive results)
Feasibility: Retention | 16 weeks
  Retention: Number of participant who continue to use SmartCP by the end of the intervention
Feasibility: Incidents | 16 weeks
  Number of adverse events reported by patients
Feasibility: User statistics | 16 weeks
  Minutes per day spent on the app during the intervention period
Feasibility: User statistics | 16 weeks
  Number per day of unique log-ins to the app during the intervention period

SECONDARY OUTCOMES:
Occurrence of crisis events: Crisis phone-calls | 16 weeks
  Number of crisis phone-calls per day to Tallaght University Hospital Advanced Nurse Practitioner
Occurrence of crisis events: Accident & Emergency | 16 weeks
  Number of attendances per week at Accident & Emergency Room in any hospital
Occurrence of crisis events: Urgent clinic | 16 weeks
  Number of urgent out-patient clinic attendances per week in Tallaght university Hospital
Symptoms: The nature and frequency of each symptom recorded using the daily symptoms tracker while using the app | 16 weeks
  Recording of tiredness or lack of energy, steatorrhoea, loss of appetite, nausea, vomiting, dyspepsia, bloating or stomach distention, excess wind or flatulence - all according to the following scale: none, mild, moderate, severe
Symptoms: Number of Alerts created by the app | 16 weeks
  The number of alerts created by the app in response to escalating symptoms requiring a phone-call or clinic attendance
Symptoms: Number of Red-Flag alerts created by the app | 16 weeks
  The number of Red-flag alerts for possible new pancreatic cancer symptoms; red-flag alert for possible new diabetes symptoms
Quality of life (QoL): Short Form-12 | 16 weeks
  Change in QoL scores measured by Short Form-12; Scores range from 0-100, with higher scores indicating better QoL
Quality of life (QoL): EQ-5D | 16 weeks
  Changes in QoL measured by EQ-5D, a self-reported questionnaire that describes a respondent's health using a descriptive system comprised of five items, each representing a different health dimension (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each dimension, respondents state whether they have no problems, slight problems, moderate problems, severe problems, or are unable to perform the activity. Score range is 0-100. Higher scores indicate better QoL
Hospitalisation: Number of admissions | 16 weeks
  Number of admissions to any hospital during the intervention period
Hospitalisation: Length of hospital stay | 16 weeks
  Length of hospital stay at any hospital during the intervention period
Use of communications features: Number of times per week patients use app communications features | 16 weeks
  Number of times per week that patients use the communication features on app (messaging the Advanced Nurse Practitioner via the app with a query)
Use of educational features: Number of times per week patients view app educational/informational features | 16 weeks
  Number of times per week patients view various videos, graphic videos, read educational texts, click on new education features provided

CONTACTS AND LOCATIONS:
Locations (1):
- University of Dublin, Trinity College, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
To be decided
Supporting Information: Study Protocol, CSR
Time Frame: After publication and for the statutory GDPR period